CLINICAL TRIAL: NCT06068595
Title: The Contribution of Targeted Musculoskeletal Ultrasound to the General Practitioner's Overall Decision-making Strategy for Patients With Suspected Musculoskeletal Pathology: a Before/After Study
Brief Title: Evaluation of the Contribution of Musculoskeletal Ultrasound to the General Practitioner's Overall Decision-making Strategy
Acronym: ECHOSTEOM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: University of Lorraine (Other)
Responsible Party: Principal Investigator, GASS Boris, Principal Investigator, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-A01995-40
Record Dates: First submitted 2023-09-22; First posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: Musculoskeletal; Anomaly
Keywords: musculoskeletal anomaly; ultrasonography; general practitioners
MeSH Terms: conditions — Musculoskeletal Abnormalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Other): Patient with musculoskeletal anomalies
  Interventions: Other: musculoskeletal ultrasound

INTERVENTIONS:
Other: musculoskeletal ultrasound — After clinical examination and medical interrogation, The investigating physician gives her decisions in the e-CRF according to the 5 axes: diagnosis (I), therapy (II), patient referral (III), prescription of additional tests (IV) and follow-up (V). The investigator performs the targeted musculoskeletal ultrasound with his personal ultrasound machine, following his usual operating procedure and give/keep the final diagnostic.

SUMMARY:
The hypothesis of this study is that musculoskeletal point of care ultrasonography would support the GP's decision and ultimately improve patient management.

The aim of this study is to evaluate, in the context of suspected musculoskeletal abnormality, the contribution of musculoskeletal point of care ultrasonography to the general practitioner's overall decision-making strategy, defined according to the following 5 axes: diagnosis (I), therapy (II), patient orientation (III), prescription of complementary examinations (IV) and follow-up (V).

DETAILED DESCRIPTION:
The study circuit takes place in a single visit.

1. The investigating physician suspects a musculoskeletal anomaly following an initial clinical examination.
2. The patient (who meets the inclusion criteria and has no non-inclusion criteria) gives consent to participate, after receiving information about the study.
3. The investigator fills in the e-CRF (appendix III), clinical examination, medical interrogation and his or her decisions according to the 5 axes, which cannot be modified, as the structure of the e-CRF planned in advance does not allow backtracking. The investigator performs the targeted musculoskeletal ultrasound with his or her personal ultrasound machine, following his or her usual operating procedure.
4. The investigator fills in the e-CRF with the results of the targeted ultrasound scan and indicates any modifications to the decision axes.

ELIGIBILITY:
Inclusion Criteria:

* Person who has received full information on the organization of the research and has given his/her consent
* Be over 18 years of age
* Present a symptomatology leading to suspicion of musculoskeletal pathology
* Be able to give consent
* Be affiliated to a social security scheme or benefit from such a scheme

Exclusion Criteria:

* Chronic inflammatory rheumatism (rheumatoid arthritis, spondylitis, psoriatic arthritis, rheumatoid pseudo-polyarthritis, juvenile idiopathic arthritis, lupus, etc.).
* Subjects benefiting from a legal protection measure (guardianship, curatorship, safeguard of justice).
* Persons deprived of their liberty by judicial or administrative decision, persons under psychiatric care under articles L3212-1 and L3213-1.
* Pregnant women
* Nursing mothers

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients | 3 years
  Percentage of patients for whom the musculoskeletal point of care ultrasonography led to a change in the GP's overall decision-making strategy (binary yes/no variable) of patients for whom led to a change in the GP's overall decision-making strategy (binary yes/no variable)

SECONDARY OUTCOMES:
Frequency of the anatomical sites | 3 years
  Frequency of the different anatomical sites (shoulder, elbow, arm, etc.) and structures (osteoarticular pathologies, tendon and retinacular pathologies, etc.) concerned
Frequency of modifications | 3 years
  Frequency of different modifications for each axis and within each axis
Frequency of diagnoses of post-CTA confirmation | 3 years
  List and frequency of diagnoses in the case of post-CTA confirmation
Frequency of diagnoses of post-CTA modifications | 3 years
  List and frequency of diagnoses in the case of post-CTA modifications
Frequency of incidental diagnoses discovered at CTA | 3 years
  Frequency and description of incidental diagnoses discovered at CTA
Frequency of modifications per patient | 3 years
  Frequency of different modifications for each axis and within each axis per patient
Calculation of the cost | 3 years
  Calculation of the cost before and after CTA estimated a posteriori on the basis of the consultation rate
Rates for the examinations and therapies | 3 years
  the rates for the examinations and therapies described
Frequency with which CTA | 3 years
  For each doctor: the frequency with which CTA is carried out in his professional practice
Time taken to carry out the CTA | 3 years
  For each doctor: the time taken to carry out the CTA
Average number of ultrasound prints | 3 years
  For each doctor: the average number of ultrasound image prints
Time taken to produce an CTA report | 3 years
  For each doctor: the time taken to produce an CTA report

CONTACTS AND LOCATIONS:
Overall Officials: Boris Gass, Pr, Principal Investigator — Central Hospital, Nancy, France
Locations (1):
- Central Hospital, Nancy, Vandoeuvre Lès Nancy, France

REFERENCES:
- [Background] Sorensen B, Hunskaar S. Point-of-care ultrasound in primary care: a systematic review of generalist performed point-of-care ultrasound in unselected populations. Ultrasound J. 2019 Nov 19;11(1):31. doi: 10.1186/s13089-019-0145-4. PMID 31749019
- [Background] Meyer R, Lin C, Yenokyan G, Ellen M. Diagnostic Utility of Ultrasound Versus Physical Examination in Assessing Knee Effusions: A Systematic Review and Meta-analysis. J Ultrasound Med. 2022 Jan;41(1):17-31. doi: 10.1002/jum.15676. Epub 2021 Mar 5. PMID 33675099
- [Background] Nazarian LN. The top 10 reasons musculoskeletal sonography is an important complementary or alternative technique to MRI. AJR Am J Roentgenol. 2008 Jun;190(6):1621-6. doi: 10.2214/AJR.07.3385. PMID 18492916
- [Background] Narula J, Chandrashekhar Y, Braunwald E. Time to Add a Fifth Pillar to Bedside Physical Examination: Inspection, Palpation, Percussion, Auscultation, and Insonation. JAMA Cardiol. 2018 Apr 1;3(4):346-350. doi: 10.1001/jamacardio.2018.0001. PMID 29490335
- [Background] Andersen CA, Davidsen AS, Brodersen J, Graumann O, Jensen MB. Danish general practitioners have found their own way of using point-of-care ultrasonography in primary care: a qualitative study. BMC Fam Pract. 2019 Jun 28;20(1):89. doi: 10.1186/s12875-019-0984-x. PMID 31253102